CLINICAL TRIAL: NCT06416267
Title: Immune Biomarkers, Genetic Risk, and the Clinical Consequences of Low Count Monoclonal B-cell Lymphocytosis (LC MBL)
Brief Title: Risk and Clinical Consequences of Low Count Monoclonal B-cell Lymphocytosis (LC MBL)
Acronym: MBL RiskConseq
Status: Not yet recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other); Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Geffen Kleinstern, Senior Lecturer, University of Haifa
Other Study IDs: MBL_RiskCons
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Monoclonal B-Cell Lymphocytosis; Chronic Lymphocytic Leukemia; Infections; Cancers; Cardiovascular Diseases; Alzheimer Disease; Dementia; Autoimmune Diseases; Parkinson Disease
Keywords: Monoclonal B cell Lymphocytosis; Genetic Risk; Outcomes; Infections; Cancers; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Infections; Neoplasms; Cardiovascular Diseases; Alzheimer Disease; Dementia; Autoimmune Diseases; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clalit Health Services: Individuals over the age of 40 attending to the Clalit HMO clinics in the North of Israel for regular blood tests.

SUMMARY:
The aim of this proposal is to identify immune biomarkers, genetic risk, and the clinical consequences of low count monoclonal B-cell lymphocytosis (LC MBL), a common premalignant condition affecting up to 17% of European adults age>40. LC MBL is a precursor to chronic lymphocytic leukemia (CLL), characterized by a circulating population of clonal B-cells. It is relatively understudied, despite emerging evidence of clinical consequences such as increased risk for life-threatening infections and lymphoid malignancies. Studies reported that male sex, age, family history of CLL, and CLL-susceptibility genetic loci were associated with LC MBL risk. These findings were reported in European ancestry individuals and have not been generalized to other thnicities. This study will provide this missing knowledge using a unique multi-ethnic Israeli population of Jews and Arabs that have one of the highest and lowest age-standardized incidence rates of CLL in the world, respectively, and characterized with different genetic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age pf 40

Exclusion Criteria:

* Individuals with lymphoproliferative disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Jewish and Arab individuals over the age of 40 attending to the Clalit HMO clinics in the North of Israel for regular blood tests
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Assess the relationship between LC MBL and life-threatening infections, hematologic malignancies, and solid tumors among Jews and Arabs in Israel | From enrollment and 15 years of follow up
  Blood samples will be screened for MBL using flow cytometry, while data on the various outcomes will be collected from electronic medical records from Clalit Health Services.
Assess the relationship between LC MBL and cardiovascular diseases, autoimmune conditions, and Alzheimer among Jews and Arabs in Israel | From enrollment and 15 years of follow up
  Blood samples will be screened for MBL using flow cytometry, while data on the various outcomes will be collected from electronic medical records from Clalit Health Services.
Identify germline genetic factors that are associated with LC MBL risk among Jews and Arabs in Israel | The first 5 years of the study
  DNA will be extracted from the blood sample and sequenced.
Evaluate the prevalence of LC MBL by Jews and Arabs and by sex in Israel. | The first 5 years of the study
  Blood samples will be screened for MBL using flow cytometry, ethnicity and sex will be determined using a demographic questionnaire
Identify immune biomarkers that are associated with LC MBL risk | The first 5 years of the study
  Blood sample will be screened for MBL using flow cytometry, and immune biomarkers will be screened from plasma samples.

SECONDARY OUTCOMES:
Assess the relationship between LC MBL and other clinical conditions | From enrollment and 15 years of follow up
  Other clinical conditions will be determined from electronic medical records from Clalit Health Services

IPD SHARING:
Plan to Share IPD: No